CLINICAL TRIAL: NCT03653650
Title: Autologous Platelet-rich Plasma in the Treatment of Persistent Corneal Epithelial Defects
Brief Title: Autologous Platelet-rich Plasma in the Treatment of Persistent Epithelial Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Collaborators: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Karim Mohamed-Noriega, Professor, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OF18-00003
Record Dates: First submitted 2018-08-16; First posted 2018-08-31 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Persistent Epithelial Defect
Keywords: Platelet-Rich Plasma; Persistent Epithelial Defect

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to three groups. Demographic characteristics and underlying etiologies will be identified. Subjects will undergo a general ophthalmologic evaluation (baseline) and PED size will be measured. Treatments will be administered until complete defect healing is achieved and visits will be scheduled weekly or as needed for continued ophthalmologic evaluation. After complete closure, subjects will be followed for three months with visits every 2 to 4 weeks to evaluate progress and identify recurrences.
Masking Description: Not blinded study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRP plus BCL (Experimental): Bandage contact lens (BCL) plus 1 autologous platelet-rich plasma (PRP) eye drop every 1 to 3 hours.
  Interventions: Combination Product: PRP plus BCL
- BCL plus PFL (Active Comparator): Bandage contact lens (BCL) plus 1 preservative-free lubricant (PFL) eye drop every 1 to 3 hours.
  Interventions: Combination Product: BCL plus PFL
- Eye patch plus ocular lubricant ointment (Active Comparator): Eye patch plus ocular lubricant ointment every 24 hours.
  Interventions: Combination Product: Eye patch plus ocular lubricant ointment

INTERVENTIONS:
Combination Product: PRP plus BCL — Bandage contact lens (BCL) plus 1 autologous platelet-rich plasma (PRP) eye drop every 1 to 3 hours.
  Arms: PRP plus BCL
Combination Product: BCL plus PFL — Bandage contact lens (BCL) plus 1 preservative-free lubricant (PFL) eye drop every 1 to 3 hours.
  Arms: BCL plus PFL
Combination Product: Eye patch plus ocular lubricant ointment — Eye patch plus ocular lubricant ointment every 24 hours.
  Arms: Eye patch plus ocular lubricant ointment

SUMMARY:
Persistent epithelial defects (PED) are corneal ulcers that do not heal within the first two weeks of treatment with artificial tears or ocular lubricant ointment. It is believed that this condition is the result of the loss of certain substances normally present in the tears that aid in the healing process of the cornea. When the eye is healthy, these ulcers typically heal rapidly. However, when there is an underlying disease such as diabetes, this healing process is altered and it takes longer for the ulcer to heal. Autologous platelet-rich plasma (PRP) is a substance that is obtained from the patient's own blood and it is believed this substance may replace those missing factors in the tears of patients with PED. The purpose of this investigation is to find out whether PRP combined with a bandage contact lens is better than preservative free lubricant combined with bandage contact lens or than eye patch with ocular lubricant ointment for the treatment of PED. Participants will be randomly assigned to one of the three groups and will get the treatment until the ulcer heals completely. We will count the days it takes for the PED to heal and based on that we will determine wich treatment is more effective (the treatment that takes the least days to heal will be considered the most effective). Since this disease is difficult to treat and doesn't have a gold standard treatment, usually the available treatments are not as good as we would like, therefore, the ulcer might progress even to perforation regardless of the treatment. In these cases, we will provide appropriate treatment for progressive corneal thinning and corneal perforation.

DETAILED DESCRIPTION:
Persistent epithelial defects (PED) are corneal lesions that do not heal within the first two weeks of conventional treatment (i.e. preservative-free lubricant, bandage contact lens (BCL), ocular lubricant ointment, eye patching). These defects are the result of the loss of certain lacrimal factors that maintain the integrity and homeostasis of the corneal epithelium and ocular surface. Normally, PED heal rapidly in the healthy eye. However, underlying ocular surface pathology can slow down the healing process and contribute to the persistence of the epithelial defect. Hematopoietic derivatives such as autologous platelet-rich plasma (PRP) may replace these missing components and eventually lead to complete healing in a faster and more comfortable way for the patient. The objective of this study is to determine if PRP combined with BCL is more effective than preservative-free lubricant combined with BCL or than eye patch with ocular lubricant ointment for the treatment of PED. Participants will be randomly assigned to one of the three groups and treatment will be administered until achieving complete defect closure. The effectiveness of each treatment will be measured in terms of days taken to achieve complete closure. Since PED is a complex disease that is difficult to treat, the available treatments are not very effective, therefore, PED might progress even to perforation regardless of the treatment. In this last scenario, we will provide appropriate treatment for progressive corneal thinning and corneal perforation

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent epithelial defect and at least one of the following diagnoses:

  * Recurrent corneal epithelial defect.
  * Neurotrophic corneal ulcer.
  * Neurotrophic keratopathy secondary to any disease (i.e. diabetes mellitus, infection with herpes simplex virus or herpes zoster virus, microbial keratitis sequelae, multiple sclerosis, Parkinson's disease, VII cranial nerve palsy, chemical or thermic burn sequelae, trauma, surgery, iatrogenic, chronic dry eye, rheumatic disease).

Exclusion Criteria:

* Patients diagnosed with:

  * Peripheral ulcerative keratitis, or Mooren's ulcer.
  * Active infectious keratitis and/or ulcers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Persistent epithelial defect healing time. | From the first day of treatment until the date of complete defect closure, assessed up to 3 months.
  Persistent epithelial defect healing time measured in days.

SECONDARY OUTCOMES:
Change in corneal sensitivity | Change from baseline corneal sensitivity at the date of defect closure, up to 3 months.
  Corneal sensitivity will be assessed with corneal esthesiometer Cochet-Bonnet.
Uncorrected visual acuity | Every week (or sooner, if needed) from date of randomization until the date of complete defect closure, up to 3 months.
  Uncorrected visual acuity will be assessed using Snellen cards. Measurements will be converted to LogMar values for statistical analysis.
Best corrected visual acuity | Every week (or sooner, if needed) from date of randomization until the date of complete defect closure, up to 3 months.
  Best corrected visual acuity will be assessed using Snellen cards. Measurements will be converted to LogMar values for statistical analysis.
Ocular pain | Every week (or sooner, if needed) from date of randomization until the date of complete defect closure, up to 3 months.
  Ocular pain will be assessed using the Wong-Baker Faces Pain Rating Scale. The scale ranges from 0 (no pain) to 10 (maximum pain), and includes 6 faces (visual representation), numbers, and written descriptions that represent the level of pain. The first face represents a pain score of 0 and it reads "no hurt"; the second face represents a pain score of 2 and it reads "hurts little bit"; the third face represents a pain score of 4 and it reads "hurts little more"; the fourth face represents a pain score of 6 and it reads "hurts even more"; the fifth face represents a pain score of 8 and it reads "hurts whole lot"; the last face represents a pain score of 10 and it reads "hurst worst". Lower values represent a better outcome.
Ocular surface symptoms | Every week (or sooner, if needed) from date of randomization until the date of complete defect closure, up to 3 months.
  Ocular surface symptoms as assessed by the Symptom Assessment in Dry Eye (SANDE) questionnaire. The SANDE questionnaire consists of two questions presented in visual analog scale. The first question assesses the frequency of dry eye syndrome and the scale ranges from "rarely" to "all the time" on a 100 mm line. The second question assesses the severity of dry eye syndrome and the scale ranges from "very mild" to "very severe" on a 100 mm line. Patients are asked to place a mark on the line to represent the extent of their symptoms, then the location of the marks on each line are measured from left to right in mm. The SANDE score is calculated by multiplying the frequency value times the severity value and obtaining the square root. Lower scores represent a better outcome.
Ocular surface symptoms | At date of randomization and at date of defect closure, up to 3 months.
  Ocular surface symptoms as assessed by the Ocular Surface Disease Index (OSDI). The OSDI questionnaire consists of 12 questions that assess dry eye symptoms and their effects on vision related function. The questionnaire is divided in 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients are asked to rate their responses on a 0 to 4 scale where 0 represents "none of the time", 1 "some of the time", 2 "half of the time", 3 "most of the time", and 4 "all of the time". The total score is calculated using the following formula: ([sum of scores for all questions answered x 100] / [total number of questions answered x 4]). Lower scores represent a better outcome.
Quality of life questionnaire | At date of randomization and at date of defect closure, up to 3 months.
  Quality of life as assessed by the National Eye Institute Visual Function Questionnaire (NEI VFQ-25). The NEI VFQ-25 questionnaire consists of 25 questions that assess the effect of visual impairment on the patient's quality of life. The 25-item questionnaire gives a score on a scale of 0 to 100, where 0 is the worst score and 100 is the best score. Higher scores represent a better outcome.
Frequency of adverse events, recurrences and/or treatment failure | These will be evaluated from the beginning of the treatment until three months after defect closure.
  Frequency of adverse events, recurrences and/or treatment failure will be evaluated during the ophthalmic evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Mohamed-Noriega, M.D., Principal Investigator — Departamento de Oftalmologia, Hospital Universitario Dr. Jose Eleuterio Gonzalez
Locations (1):
- Departamento de Oftalmologia, Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsubota K, Goto E, Shimmura S, Shimazaki J. Treatment of persistent corneal epithelial defect by autologous serum application. Ophthalmology. 1999 Oct;106(10):1984-9. doi: 10.1016/S0161-6420(99)90412-8. PMID 10519596
- [Background] Chen J, Chen P, Backman LJ, Zhou Q, Danielson P. Ciliary Neurotrophic Factor Promotes the Migration of Corneal Epithelial Stem/progenitor Cells by Up-regulation of MMPs through the Phosphorylation of Akt. Sci Rep. 2016 May 13;6:25870. doi: 10.1038/srep25870. PMID 27174608
- [Background] Ljubimov AV, Saghizadeh M. Progress in corneal wound healing. Prog Retin Eye Res. 2015 Nov;49:17-45. doi: 10.1016/j.preteyeres.2015.07.002. Epub 2015 Jul 18. PMID 26197361
- [Background] Nugent RB, Lee GA. Ophthalmic use of blood-derived products. Surv Ophthalmol. 2015 Sep-Oct;60(5):406-34. doi: 10.1016/j.survophthal.2015.03.003. Epub 2015 Apr 15. PMID 26077627
- [Background] Alio JL, Rodriguez AE, WrobelDudzinska D. Eye platelet-rich plasma in the treatment of ocular surface disorders. Curr Opin Ophthalmol. 2015 Jul;26(4):325-32. doi: 10.1097/ICU.0000000000000169. PMID 26058033
- [Background] Alio JL, Abad M, Artola A, Rodriguez-Prats JL, Pastor S, Ruiz-Colecha J. Use of autologous platelet-rich plasma in the treatment of dormant corneal ulcers. Ophthalmology. 2007 Jul;114(7):1286-1293.e1. doi: 10.1016/j.ophtha.2006.10.044. Epub 2007 Feb 26. PMID 17324465
- [Background] Kim KM, Shin YT, Kim HK. Effect of autologous platelet-rich plasma on persistent corneal epithelial defect after infectious keratitis. Jpn J Ophthalmol. 2012 Nov;56(6):544-50. doi: 10.1007/s10384-012-0175-y. Epub 2012 Sep 13. PMID 22972393